CLINICAL TRIAL: NCT00366561
Title: Retrospective Review of Neonates With Neurological Complications Following Cardiac Surgery
Brief Title: Neonates With Neurological Complications
Status: Completed | Type: Observational
Sponsor: Children's Healthcare of Atlanta (Other)
Responsible Party: Sponsor
Other Study IDs: 06-139
Record Dates: First submitted 2006-08-17; First posted 2006-08-21 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Congenital Disorders
Keywords: neonates; neurological complications; surgery
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this retrospective study is to identify all neonates (newborns < 30 days of age) from January 1, 2002 through June 20, 2006 at Children's Healthcare of Atlanta who have suffered neurological complications following cardiac surgery. This retrospective study is important to identify the incidence, care and follow-up of neurological complications at this institution

DETAILED DESCRIPTION:
Studies have shown that between one-quarter and one-half of infants undergoing cardiac surgery will suffer brain injury during surgery (the perioperative period). Some infants with congenital heart disease have neurological injury prior to cardiac surgery as a result of cyanosis, acidosis and abnormal circulation. The spectrum of neurological injury ranges from agitation and subtle disturbances in learning and new memory acquisition to visual and motor development abnormalities, seizures, stroke and encephalopathy.

The patient will be identified from the cardiothoracic surgery database. Their hospital medical records and the neurological database will be reviewed for type of neurological complication (i.e. seizure, stroke), neuro-imaging and any mortality for these patients. We will review the patient outcome data that is available, after the initial surgery, through June 20, 2006. No patients will be contacted.

ELIGIBILITY:
Inclusion Criteria:

* Children's Healthcare of Atlanta patients
* January 1, 2002 through June 20, 2006
* < 30 days of age
* neurological complications following cardiac surgery

Exclusion Criteria:

* Those who do not meet inclusion criteria

Max Age: 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All neonates (newborns < 30 days of age) from January 1, 2002 through June 20, 2006 at Children's Healthcare of Atlanta who have suffered neurological complications following cardiac surgery.
Sampling Method: Non-Probability Sample
Enrollment: 810 (Actual)
Dates: Start 2002-01; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
The purpose of this study was to examine short term outcomes following cardiac surgery in premature neonates. | 6 years
  In congenital cardiac defects where there was a choice of palliation vs complete anatomic repair, premature neonates underwent palliative procedures more frequently than term neonates. Premature neonates spent more days of mechanical ventilation compared to their term counterparts. Importantly, there was no difference in mortality between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Janet M Simsic, MD, Principal Investigator — Sibley Heart Center Cardiology at Children's Healthcare of Atlanta
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States